CLINICAL TRIAL: NCT07210411
Title: Acute and Chronic Repercussion of Spinal Cord Stimulation After Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ryan J. Solinsky, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-001000
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Experimental): Control participants without a spinal cord injury
  Interventions: Diagnostic Test: Tests of sympathetic inhibition; Diagnostic Test: Tests of above level sympathetic activation; Diagnostic Test: Testing of below level sympathetic activation
- Transcutaneous stimulation (Experimental): Individuals with spinal cord injury receiving transcutaneous stimulation
  Interventions: Diagnostic Test: Tests of sympathetic inhibition; Diagnostic Test: Tests of above level sympathetic activation; Diagnostic Test: Testing of below level sympathetic activation; Device: Transcutaneous stimulation
- Epidural stimulation (Experimental): Individuals with spinal cord injury receiving epidural stimulation
  Interventions: Diagnostic Test: Tests of sympathetic inhibition; Diagnostic Test: Tests of above level sympathetic activation; Diagnostic Test: Testing of below level sympathetic activation; Device: Epidural stimulation

INTERVENTIONS:
Diagnostic Test: Tests of sympathetic inhibition — Bolus phenylephrine infusion using the Oxford technique will generate the need to inhibit sympathetic activity. Similarly, resting state Mayer waves will be assessed with regard to heart rate and blood pressure responses.
Diagnostic Test: Tests of above level sympathetic activation — Cold pressor test of the hand will be used to cause sympathetic activation. Valsalva's maneuver will assess the ability to buffer against blood pressure fall (phase II).
Diagnostic Test: Testing of below level sympathetic activation — Cold pressor test of the foot and bladder pressor response (in individuals with SCI) will be tested.
Device: Epidural stimulation — Currently implanted epidural stimulation will be used during diagnostic testing.
  Arms: Epidural stimulation
Device: Transcutaneous stimulation — Transcutaneous stimulation will be used for participants with spinal cord injury without an implanted stimulator during diagnostic testing.
  Arms: Transcutaneous stimulation

SUMMARY:
The purpose of this research is to learn about how the participant's body is able to balance changes in blood pressure, and how spinal cord stimulation affects these changes as well as immune & cardiovascular function in participants with spinal cord injury.

ELIGIBILITY:
Inclusion criteria

* Age 18-50.
* American Spinal Injury Association Impairment Scale A-D,64 to encompass a representational spectrum of autonomic dysfunction after spinal cord injury.
* Neurological level of injury, C6-T8, as defined by the International Standards for Neurological Classification of Spinal Cord Injury.64 Incorporating level of injury over this broad range to capture the spectrum of autonomic dysfunction. Individuals with injuries below T8 will not be included to ensure transcutaneous spinal cord stimulation does not occur over the injury/glial scar, where it may have altered properties. The C6 level was chosen to ensure hand cold pressor stimuli triggers above level sympathetic activation.
* Time since injury of greater than six months, given early changes in spinal cord connectivity and recovery prior to this.
* Both individuals with and without currently implanted epidural spinal cord stimulators will be enrolled.
* Twenty uninjured controls will also be enrolled.

Exclusion criteria

* History of clinically diagnosed cardiovascular disease, diabetes, autonomic neuropathies, neurological disorders (with exception of spinal cord injury for individuals in those cohorts), or are active smokers.
* Individuals who are taking betablockers, antihypertensives, or other sympathetically active medications which they are unable to hold.
* Women who are pregnant or lactating, given known hormonal influences on autonomic regulation.65,66
* Cognitive issues preventing informed consent for participation.
* Body mass index >30 kg/m2 for the uninjured controls only given increased risk of prediabetes and potential confounding normative values.
* taking or being administered a medication known to potentially have adverse interactions with phenylephrine
* in the judgement of the principal investigator, any illness or condition that will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-04-01 (Estimated)

PRIMARY OUTCOMES:
Valsalva Maneuver Phase II | During laboratory diagnostic testing session
  Presence or absence of phase II on Valsalva maneuver testing, which takes approximately 15 seconds to complete. This will be repeated x3.

SECONDARY OUTCOMES:
Beat-to-beat heart rate | During laboratory diagnostic testing session
  Electrocardiogram will record continuous measures with changes in R-R interval (ms) quantified and compared to baseline.
Beat-to-beat blood pressure | During laboratory diagnostic testing session
  Non-invasive continuous blood pressure monitors will be used, with changes in systolic and diastolic pressure (in mmHg) from resting baseline measured.
Continuous galvanic skin response | During laboratory diagnostic testing session
  Changes from resting state conductance with be quantified with a smartwatch.
Quantify autonomic dysreflexia and orthostatic hypotension | Baseline, prior to laboratory diagnostic testing session
  Participants will be given the Autonomic Dysfunction Following Spinal Cord Injury questionnaire (score range 0-436, with higher scores indicating more autonomic dysfunction).
Respiration | During laboratory diagnostic testing session
  Elastic respiratory transducer bands around mid-chest and upper abdomen will monitor breathing depth and frequency.
Beat-by-Beat Popliteal and Brachial Blood Flow | During laboratory diagnostic testing session
  The investigators will use Doppler derived flow velocities to estimate whole limb blood flow through the popliteal and brachial arteries
Immunology Blood Draw | During laboratory diagnostic testing session
  Baseline samples will be collected and compared against changes to blood pressure.
Serum Catecholamines and Cortisol | During laboratory diagnostic testing session
  Baseline resting catecholamines (norepinephrine, epinephrine, dopamine) and cortisol will be drawn from the IV after 10 minutes of quiet rest at baseline and prior to bladder filling or foot cold pressor. Just prior to the conclusion of this testing, an additional blood draw will take place through the IV to assess changes in these levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Solinsky, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Solinsky R, Burns K, Tuthill C, Hamner JW, Taylor JA. Transcutaneous spinal cord stimulation and its impact on cardiovascular autonomic regulation after spinal cord injury. Am J Physiol Heart Circ Physiol. 2024 Jan 1;326(1):H116-H122. doi: 10.1152/ajpheart.00588.2023. Epub 2023 Nov 10. PMID 37947438
- [Background] Solinsky R, Burns K, Hamner JW, Veith DD, Singer W, Taylor JA. A Novel Testing Battery for Preserved Autonomic Regulation Following Spinal Cord Injury and New Translationally Focused Data Representation. Top Spinal Cord Inj Rehabil. 2025 Spring;31(2):50-61. doi: 10.46292/sci24-00071. Epub 2025 Jun 19. PMID 40585014